CLINICAL TRIAL: NCT04962438
Title: Effects of Anti-VEGF Targeted Drugs on Patients' Blood Pressure and Endothelial Function
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Cardiac safety
Record Dates: First submitted 2021-06-27; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Cardiac Toxicity; VEGF; Endothelial Dysfunction
Keywords: Cardiac safety; anti-VEGF drugs; Endothelial dysfunction
MeSH Terms: conditions — Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tumor patients using anti-VEGF drugs
  Interventions: Drug: Anti-VEGF

INTERVENTIONS:
Drug: Anti-VEGF — Anti-tumor drugs targeting the vascular endothelial growth factor (VEGF) signaling pathway

SUMMARY:
Explore the effects of anti-VEGF targeted drugs on blood pressure and endothelial function in cancer patients.

DETAILED DESCRIPTION:
Thirty tumor patients with anti-VEGF drugs were selected. Demographic information and clinical information of all patients were collected before chemotherapy. Ambulatory blood pressure monitoring and endothelial function measurement (PWV, EndoPAT) were performed. Ambulatory blood pressure and PWV were reviewed at 2 weeks and 1 month. And EndoPAT, to evaluate the effects of anti-VEGF drugs on blood pressure and endothelial function in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Tumor patients using anti-VEGF drugs

Exclusion Criteria:

* Hypertension, coronary heart disease, valvular heart disease, cardiomyopathy and other organic heart diseases, exclude liver and kidney failure, severe cerebrovascular disease, chronic obstructive pulmonary disease, rheumatic immune system disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Thirty tumor patients selected for anti-VEGF drugs, demographic and clinical information of all patients were collected before chemotherapy, ambulatory blood pressure monitoring, endothelial function determination (PWV, EndoPAT)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-07-05 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Time ending | 1 month
  30 days after using the Anti-VEGF Targeted Drugs

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided